CLINICAL TRIAL: NCT06382142
Title: A Phase III Randomized Controlled Clinical Study Comparing BL-B01D1 With Chemotherapy of Physician's Choice in Patients With Unresectable Locally Advanced or Metastatic Triple-Negative Breast Cancer After Taxane Failure
Brief Title: A Study Comparing BL-B01D1 With Chemotherapy of Physician's Choice in Patients With Unresectable Locally Advanced or Metastatic Triple-Negative Breast Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BL-B01D1-307
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Triple-Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — eribulin; Vinorelbine; Gemcitabine; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BL-B01D1 (Experimental): Participants receive BL-B01D1 as intravenous infusion for the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-B01D1
- Eribulin or Vinorelbine or Gemcitabine or Capecitabine (Experimental): Participants receive Eribulin or Vinorelbine or Gemcitabine or Capecitabine in the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: Eribulin; Drug: Vinorelbine; Drug: Gemcitabine; Drug: Capecitabine

INTERVENTIONS:
Drug: BL-B01D1 — Administration by intravenous infusion for a cycle of 3 weeks.
  Other Names: iza-bren; izalontamab brengitecan; BMS-986507
  Arms: BL-B01D1
Drug: Eribulin — Administration by intravenous bolus for a cycle of 3 weeks.
  Arms: Eribulin or Vinorelbine or Gemcitabine or Capecitabine
Drug: Vinorelbine — Administration by intravenous infusion for a cycle of 3 weeks.
  Arms: Eribulin or Vinorelbine or Gemcitabine or Capecitabine
Drug: Gemcitabine — Administration by intravenous infusion for a cycle of 3 weeks.
  Arms: Eribulin or Vinorelbine or Gemcitabine or Capecitabine
Drug: Capecitabine — Oral administration for a cycle of 3 weeks.
  Arms: Eribulin or Vinorelbine or Gemcitabine or Capecitabine

SUMMARY:
This trial is a registered phase III, randomized, open-label, multicenter study designed to evaluate the efficacy and safety of BL-B01D1 in patients with unresectable locally advanced or metastatic Triple-Negative breast cancer after taxane failure.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent and follow the requirements of the protocol;
2. No gender limit;
3. Age ≥18 years old and ≤75 years old;
4. Expected survival time ≥3 months;
5. Patients with unresectable, locally advanced or metastatic triple-negative breast cancer;
6. Consent to provide archival tumor tissue samples or fresh tissue samples of primary or metastatic lesions within 3 years;
7. The subjects had received 1-2 lines of chemotherapy regimens in the locally advanced or metastatic stage, and had been treated with taxanes previously;
8. Acceptability of chemotherapy with eribulin, capecitabine, gemcitabine, or vinorelbine, as assessed by the investigator;
9. Patients with baseline brain metastases should have received treatment for all brain metastases and be stable;
10. Must have at least one measurable lesion that meets the RECIST v1.1 definition;
11. ECOG score 0 or 1;
12. Toxicity of previous antineoplastic therapy has returned to ≤ grade 1 defined by NCI-CTCAE v5.0;
13. No severe cardiac dysfunction, left ventricular ejection fraction ≥50%;
14. No blood transfusion, no use of cell growth factors and/or platelet raising drugs within 14 days before the first use of the study drug, and the organ function level must meet the requirements;
15. Coagulation function: international normalized ratio ≤1.5, and activated partial thromboplastin time ≤1.5×ULN;
16. Urine protein ≤2+ or < 1000mg/24h;
17. For premenopausal women with childbearing potential, a pregnancy test must be performed within 7 days before the initiation of treatment, serum pregnancy must be negative, and must be non-lactating; All enrolled patients (male or female) were advised to use adequate barrier contraception throughout the treatment cycle and for 6 months after the end of treatment.

Exclusion Criteria:

1. Prior receipt of an ADC with a TOPI inhibitor as a toxin;
2. Prior receipt of an ADC or antibody drug targeting EGFR and/or HER3;
3. Chemotherapy, biological therapy, immunotherapy, etc. within 4 weeks or 5 half-lives before the first dose, small molecule targeted therapy within 5 days, palliative radiotherapy and anti-tumor therapy within 2 weeks;
4. Anthracycline equivalent cumulative dose of adriamycin > 360 mg/m2;
5. History of severe cardiovascular or cerebrovascular disease;
6. Unstable thrombotic events requiring therapeutic intervention within 6 months before screening;
7. QT prolongation, complete left bundle branch block, III degree atrioventricular block, frequent and uncontrollable arrhythmia;
8. Active malignancy diagnosed within 5 years before randomization;
9. Hypertension poorly controlled by two antihypertensive drugs;
10. Patients with poor blood glucose control before the first dose;
11. A history of interstitial lung disease requiring steroid therapy, or current radiation pneumonitis, or a suspicion of such disease;
12. Complicated with pulmonary diseases leading to clinically severe respiratory impairment;
13. Patients with carcinomatous meningitis (meningeal metastasis) or brain stem metastasis or spinal cord compression;
14. Have a history of allergy to recombinant humanized antibodies or any of the ingredients of BL-B01D1;
15. A history of autologous or allogeneic stem cell transplantation;
16. Human immunodeficiency virus antibody positive, active hepatitis B virus infection, or hepatitis C virus infection;
17. Severe infection within 4 weeks before randomization; Evidence of pulmonary infection or active pulmonary inflammation within 2 weeks before randomization;
18. Patients with massive or symptomatic effusions or poorly controlled effusions;
19. Imaging examination showed that the tumor had invaded or enveloped the large blood vessels in the abdomen, chest, neck, and pharynx;
20. Were receiving long-term systemic corticosteroids or equivalent active anti-inflammatory drugs or any form of immunosuppressive therapy before randomization;
21. Received other unmarketed investigational drug or treatment within 4 weeks before the first dose;
22. Patients with superior vena cava syndrome should not be rehydrated;
23. A history of severe neurological or mental illness;
24. Severe unhealed wound, ulcer, or fracture within 4 weeks before signing the informed consent;
25. Subjects with clinically significant bleeding or obvious bleeding tendency within 4 weeks before signing the informed consent;
26. History of intestinal obstruction, inflammatory bowel disease, or extensive bowel resection or presence of Crohn's disease, ulcerative colitis, or chronic diarrhea;
27. Patients scheduled for vaccination or receiving live vaccine within 28 days before the first dose;
28. Other circumstances that were assessed by the investigator as inappropriate for participation in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2024-06-21 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 24 months
  Progression-free survival (PFS) as assessed by BIRC is defined as the time between the date subjects are randomized and the first observation of disease progression (based on BICR's image-based assessment) or death.
Overall survival (OS) | Up to approximately 24 months
  Overall survival (OS) is defined as the time between the subject's randomization date and subject's death.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 24 months
  Objective response rate (ORR) is defined as the number of CR and PR in the treatment and control groups divided by the number of that group in the full analysis set (FAS).
Disease Control Rate (DCR) | Up to approximately 24 months
  Disease Control Rate (DCR) : Percentage of all randomized subjects who rated the best overall response (BOR) as complete response (CR), partial response (PR), and disease stabilization (SD) according to RECIST 1.1 criteria.
Duration of Response (DOR) | Up to approximately 24 months
  Duration of Response (DOR) : defined as the period from the date when tumor response is first recorded to the date when objective tumor progression is first recorded or the date of death.
Treatment Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-B01D1. The type, frequency and severity of TEAE will be evaluated during the treatment of BL-B01D1.
Anti-drug antibody (ADA) | Up to approximately 24 months
  Frequency of anti-BL-B01D1 antibody (ADA) will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Jiong Wu, Principal Investigator — Fudan University; Jian Zhang, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China